CLINICAL TRIAL: NCT00244374
Title: A Randomized Trial of Vaccine Adherence in Young IDU
Brief Title: A Randomized Trial of Vaccine Adherence in Young Injection Drug Users
Acronym: UFO VAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: NIDA-17476-1; R01DA017476 (NIH)
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-07

CONDITIONS: Medication Adherence; Substance Abuse, Intravenous; Risk Behavior; Hepatitis A; Hepatitis B; Hepatitis C
MeSH Terms: conditions — Medication Adherence; Substance Abuse, Intravenous; Risk-Taking; Hepatitis A; Hepatitis B; Hepatitis C | interventions — twinrix; Engerix-B; Community-Institutional Relations; Needle-Exchange Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- AIC, Hepatitis A & B vaccine (Experimental): Subjects randomized to a public health department clinic, the Adult Immunization Clinic (AIC), for administration of viral hepatitis immunizations at Month 1, 2, 6.
  Interventions: Biological: Hepatitis A & B vaccine; Behavioral: AIC
- AIC, Outreach, Hepatitis A & B vaccine (Experimental): AIC + outreach: Subjects randomized to a public health department clinic, the Adult Immunization Clinic (AIC)) for administration of viral hepatitis immunizations at Month 1, 2, 6, plus outreach worker adherence support to receive all immunizations
  Interventions: Biological: Hepatitis A & B vaccine; Behavioral: Outreach; Behavioral: AIC
- SEP, Hepatitis A & B vaccine (Experimental): SEP only: Subjects randomized to a set of syringe exchange programs for administration of viral hepatitis immunizations at Month 1, 2, 6.
  Interventions: Biological: Hepatitis A & B vaccine; Behavioral: SEP
- SEP, Outreach, Hepatitis A & B vaccine (Experimental): Subjects randomized to a set of syringe exchange programs for administration of viral hepatitis immunizations at Month 1, 2, 6, plus outreach worker adherence support to receive all immunizations
  Interventions: Biological: Hepatitis A & B vaccine; Behavioral: Outreach; Behavioral: SEP

INTERVENTIONS:
Biological: Hepatitis A & B vaccine — Each subject will receive a total of 4 immunizations over 6 months on a 0-1-2-6 month schedule. At the initial visit, subjects>18 years of age will receive the Twinrix vaccine and subjects<18 years of age will receive the Engerix-B vaccine. Cohort subjects>18 years found to have HAV antibody at screening will receive Engerix-B for their remaining 3 immunizations. All subjects will receive: an immunization record with the first vaccine dose entered and the dates the next doses are due; helpful hints for remembering vaccine appointments; and written instructions on where and how to get immunized outside of SF.
  Other Names: Twinrix; Engerix-B
Behavioral: Outreach — Outreach worker vaccine adherence support: Half of cohort subjects will be assigned to outreach worker vaccine adherence support and will meet with their outreach workers from Haight Ashbury Youth Outreach Team (HAYOT) and Glide Health Services on the day of vaccine cohort study enrollment. Intensive vaccination tracking and in-person outreach support will begin one week before the second and third vaccine doses are due, and again two weeks before the fourth dose is due.
  Other Names: Haight Ashbury Youth Outreach Team (HAYOT); Glide Health Services
  Arms: AIC, Outreach, Hepatitis A & B vaccine; SEP, Outreach, Hepatitis A & B vaccine
Behavioral: AIC — The Adult Immunization Clinic (AIC) is a public low-cost vaccine clinic located centrally at 101 Grove Street in the lobby of the San Francisco Department of Public Health (SFDPH). The clinic is open from Monday-Friday 9 a.m. to 4 p.m. Nurses at the AIC will be available 40 hours/week to administer free immunizations to study subjects.
  Other Names: Adult Immunization Clinic (AIC); San Francisco Department of Public Health (SFDPH)
  Arms: AIC, Hepatitis A & B vaccine; AIC, Outreach, Hepatitis A & B vaccine
Behavioral: SEP — Subjects randomized to a set of syringe exchange programs for administration of viral hepatitis immunizations at Month 1, 2, 6. Research nurses will provide 16 hours/week of vaccine administration services at SEPs well attended by young IDU. The San Francisco Needle Exchange (SFNE) serves primarily youth and young adults on Mondays, Wednesdays, and Fridays from 5-7 p.m. in an indoor location in the Haight-Ashbury district. A study nurse will be at SFNE for a total of 6 hours per week. HIV Prevention Project (HPP) sites also operate for 2 hrs each (Tues, Thu, Fri, Sat). Medical services are provided either in a clinic setting at indoor sites (6th Street) or at outdoor sites (Hemlock Alley, Duboce). A study nurse will attend each of these 5 weekly sites for a total of 10 hours/week.
  Other Names: syringe exchange; needle exchange; harm reduction; San Francisco Needle Exchange (SFNE); HIV Prevention Project (HPP)
  Arms: SEP, Hepatitis A & B vaccine; SEP, Outreach, Hepatitis A & B vaccine

SUMMARY:
The purpose of this study is to compare the effects of (a) immunization setting and (b) outreach worker support on young injection drug users' (IDU) adherence to a multiple dose immunization schedule with a combined hepatitis A virus (HAV) inactivated and hepatitis B virus (HBV) recombinant vaccine.

DETAILED DESCRIPTION:
This is a research trial consisting of a cross-sectional screening study and a prospective cohort study (randomized, 2x2 factorial design). The primary aim of the study is to evaluate the effects of immunization setting and outreach worker support on young IDU's adherence to a multiple dose immunization schedule with a combined HAV and HBV vaccine. Secondarily, the study will 1) explore the feasibility of a remote immunization network and web-based vaccine registry to improve immunization coverage of transient young IDU, 2) examine the effect of hepatitis C virus (HCV) infection in vaccine effectiveness, and 3) assess behavior change and vaccine attitudes in young IDU participating in a preventive vaccine trial.

Subjects in the screening study complete an interview, receive counseling and testing for HIV, HAV, HBV and HCV, and return in one week for test results and risk reduction counseling. Subjects eligible for the cohort study receive their first immunizations at enrollment and then are randomized to receive subsequent vaccines at either a set of syringe exchange programs (SEP) or at a public health adult immunization clinic (AIC). Subjects also are randomized to receive vaccine reminders from an outreach worker or no outreach worker support. Each subject receives a total of 4 immunizations over 6 months. Follow up visits include interviews, counseling, and viral testing. Study participation is for 12 months.

ELIGIBILITY:
Inclusion Criteria (screening study):

* age 14-29 at screening
* injected drugs in the prior 30 days

Exclusion Criteria (screening study):

* Prior positive HIV antibody test
* Prior HBV immunization

Inclusion Criteria (vaccine cohort):

* participated in the screening study
* tested negative for HIV-1 antibody and HBV markers in the screening study
* returned for screening test results within 30 days of testing

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 546 (Actual)
Dates: Start 2004-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula J Lum, M.D., M.P.H., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Medical Cen, San Francisco, California, United States

REFERENCES:
- [Result] Hahn JA, Page-Shafer K, Ford J, Paciorek A, Lum PJ. Traveling young injection drug users at high risk for acquisition and transmission of viral infections. Drug Alcohol Depend. 2008 Jan 11;93(1-2):43-50. doi: 10.1016/j.drugalcdep.2007.08.016. Epub 2007 Nov 5. PMID 17980513
- [Result] Etcheverry MF, Lum PJ, Evans JL, Sanchez E, de Lazzari E, Mendez-Arancibia E, Sierra E, Gatell JM, Page K, Joseph J. HIV vaccine trial willingness among injection and non-injection drug users in two urban centres, Barcelona and San Francisco. Vaccine. 2011 Feb 24;29(10):1991-6. doi: 10.1016/j.vaccine.2010.12.043. Epub 2011 Jan 15. PMID 21241735
- [Result] Lum PJ, Hahn JA, Shafer KP, Evans JL, Davidson PJ, Stein E, Moss AR. Hepatitis B virus infection and immunization status in a new generation of injection drug users in San Francisco. J Viral Hepat. 2008 Mar;15(3):229-36. doi: 10.1111/j.1365-2893.2007.00933.x. PMID 18233994
- See also: The UFO Study — http://caps.ucsf.edu/resources/project-websites/ufo-study/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 08/31/2004 and 11/30/2007, street-based outreach workers distributed study invitation cards to potential subjects in neighborhoods of San Francisco where young injection drug users (IDU) are known to congregate. Initial Contact form included self-reported age, IDU in last 30 days, hepatitis B immunization and HIV-positive status.
Pre-assignment Details: 1304 persons completed initial contact form; 645 were eligible and 546 opted to participate in the cross-sectional study. The vaccine adherence cohort (n=167) included participants enrolled prior to 3/31/2007 who met additional eligibility criteria.
Groups:
- Cross-sectional/Screening: Cross-sectional screening to determine eligibility for vaccine adherence trial
- AIC Only: Subjects randomized to a public health department clinic, the Adult Immunization Clinic (AIC), for administration of viral hepatitis immunizations at Month 1, 2, 6.
- AIC + Outreach: Subjects randomized to a public health department clinic, the Adult Immunization Clinic (AIC)) for administration of viral hepatitis immunizations at Month 1, 2, 6, plus outreach worker adherence support to receive all immunizations
- SEP Only: Subjects randomized to a set of syringe exchange programs for administration of viral hepatitis immunizations at Month 1, 2, 6.
- SEP + Outreach: Subjects randomized to a set of syringe exchange programs for administration of viral hepatitis immunizations at Month 1, 2, 6, plus outreach worker adherence support to receive all immunizations
Period: Pre-Randomization Cross-sectional Study
Arm/Group | Cross-sectional/Screening | AIC Only | AIC + Outreach | SEP Only | SEP + Outreach
Started | 546 | 0 | 0 | 0 | 0
Completed | 409 | 0 | 0 | 0 | 0
Not Completed | 137 | 0 | 0 | 0 | 0
Not completed — Did not complete baseline procedures | 105 | 0 | 0 | 0 | 0
Not completed — Technical difficulty loss of data | 17 | 0 | 0 | 0 | 0
Not completed — Did not respond to willingness questions | 14 | 0 | 0 | 0 | 0
Not completed — Interviewer lack confidence in responses | 1 | 0 | 0 | 0 | 0
Period: Evaluation for Vaccine Adherence Cohort
Arm/Group | Cross-sectional/Screening | AIC Only | AIC + Outreach | SEP Only | SEP + Outreach
Started | 440 (440 study participants enrolled prior to 3/31/2007 were evaluated for vaccine adherence cohort) | 0 | 0 | 0 | 0
Eligible for Vaccine Adherence Cohort | 217 | 0 | 0 | 0 | 0
Completed | 167 | 0 | 0 | 0 | 0
Not Completed | 273 | 0 | 0 | 0 | 0
Not completed — Evidence of hepatitis B immunization | 172 | 0 | 0 | 0 | 0
Not completed — Unable/unwilling to complete enrollment | 51 | 0 | 0 | 0 | 0
Not completed — Did not return for screening test result | 34 | 0 | 0 | 0 | 0
Not completed — Returned for results after enroll window | 4 | 0 | 0 | 0 | 0
Not completed — Declined to participate in cohort | 12 | 0 | 0 | 0 | 0
Period: Vaccine Adherence Cohort
Arm/Group | Cross-sectional/Screening | AIC Only | AIC + Outreach | SEP Only | SEP + Outreach
Started | 0 (Eligible and willing cross-sectional study participants progressed to adherence cohort randomization) | 47 | 43 | 36 | 41
Completed | 0 | 47 | 43 | 36 | 41
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants in pre-randomization cross-sectional study
Arm/Group | All Participants
Number analyzed (Participants) | 546
Age, Customized [Number; unit: Participants]
  Age 0 - 14 years | 0
  Age 15 - 29 years | 546
  Age >= 30 years | 0
Sex/Gender, Customized [Number; unit: Participants] — Gender: Male, Female, Unknown or Not Reported
  Participants
    Female | 149
    Male | 395
    Unknown/Other/Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52
  Not Hispanic or Latino | 460
  Unknown or Not Reported | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 11
  White | 392
  More than one race | 63
  Unknown or Not Reported | 61
Region of Enrollment [Number; unit: participants]
  United States | 546

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Series Completion
Description: The primary outcome was the completion of the four-dose vaccine series in a 12 month period.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | AIC Only | AIC + Outreach | SEP Only | SEP + Outreach
Number analyzed (Participants) | 47 | 43 | 36 | 41
participants
  Completed 4 vaccine doses | 16 | 20 | 8 | 10
  Completed <4 vaccine doses | 31 | 23 | 28 | 31

2. Secondary Outcome: Hepatitis B Surface Antibody Seroconversion After 3 Vaccine Doses
Description: To examine the effect of hepatitis C virus (HCV) infection on vaccine effectiveness, we compared anti-HBs (antibody to the hepatitis B surface antigen) seroconversion after three vaccine doses between anti-HCV (antibody to the hepatitis C virus) positive and anti-HCV negative participants.
Time Frame: 12 months
Population: 139 participants who completed 3 vaccine doses were included in the analysis. Enrollment for this aim continued after enrollment into the 12-month vaccine adherence trial closed; an additional 51 persons were found eligible and enrolled.
Measure: Number; unit: Participants
Groups:
- Anti-HCV Positive: Participants tested positive for Hepatitis C Virus (HCV) antibody
- Anti-HCV Negative: Participants tested negative for Hepatitis C Virus (HCV) antibody
Arm/Group | Anti-HCV Positive | Anti-HCV Negative
Number analyzed (Participants) | 31 | 108
Participants
  anti-HBs positive | 20 | 90
  anti-HBs negative | 11 | 18

3. Secondary Outcome: Viral Transmission Risk Behavior Association With Travel
Description: In a cross-sectional analysis of 355 subjects enrolled between 2004 and 2006, we estimate the associations between travel in the 3 months prior to baseline and behaviors occurring in the 30 days prior to baseline, such as drug and alcohol and sexual behaviors, that may facilitate the spread of viral infections.
Time Frame: Baseline
Population: Cross-sectional analysis of 355 subjects enrolled between 2004 and 2006
Measure: Number; unit: percentage of participants
Groups:
- Traveled in the Prior 3 Months: Participants who answered "yes" when asked if they had "been on the road or traveling outside of San Francisco" in the prior 3 months, and whose last 3 travel destinations were at least 30 miles from San Francisco
- Did Not Travel in the Prior 3 Months: Participants who answered "no" when asked if they had "been on the road or traveling outside of San Francisco" in the prior 3 months, or whose last 3 travel destinations within 30 miles of San Francisco
Arm/Group | Traveled in the Prior 3 Months | Did Not Travel in the Prior 3 Months
Number analyzed (Participants) | 221 | 134
percentage of participants
  Used (injected/snorted/smoked) heroin | 83.7 | 76.1
  Used (injected/snorted/smoked) powder cocaine | 55.7 | 41.0
  Used (injected/snorted/smoked) crack cocaine | 56.5 | 45.5
  Used (injected/snorted/smoked) methamphetamine | 67.4 | 78.4
  More than one of the above (poly-substance use) | 87.2 | 76.3
  Heavy drinking (>14, >21 per week; women, men) | 52.3 | 13.7
  Drank until blacked out | 36.8 | 13.7
  Injected daily, past 30 days | 23.5 | 33.6
  Number of injecting partners >=5 | 59.7 | 41.1
  Lent a needle/syringe | 53.3 | 46.3
  Injected with someone else's used needle/syringe | 52.3 | 37.8
  Pooled money to buy drugs | 86.4 | 66.2
  Shared cooker/spoon to prepare drugs | 67.0 | 48.1
  Syringe was backloaded | 62.7 | 47.4
  Did someone's "rinse" | 42.5 | 34.3
  Median number of sexual partners >=2 | 58.4 | 38.1
  Traded sex for money or drugs | 11.3 | 11.9
  >90% condom use if sexually active | 24.3 | 22.5
Statistical Analysis 1: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p = 0.05, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.80 to 2.44] — Odds for travel in the past 3 months as a risk factor for used (injected/snorted/smoked) heroin in the past 30 days
Statistical Analysis 2: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p = 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.12 to 2.76] — Odds for travel in the past 3 months as a risk factor for having Used (injected/snorted/smoked) powder cocaine in the past 30 days
Statistical Analysis 3: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p = 0.05, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.00 to 2.44] — Odds for travel in the prior 3 months as a risk factor for having Used (injected and/or snorted) crack cocaine in the past 30 days
Statistical Analysis 4: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p = 0.03, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.35 to 0.98] — Odds for travel in the prior 3 months as a risk factor for having Used (injected/snorted/smoked) methamphetamine in the past 30 days
Statistical Analysis 5: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.11 to 3.59] — Odds for travel in the prior 3 months as a risk factor for poly-substance use in the past 30 days
Statistical Analysis 6: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 6.87, 95% CI 2-sided [3.84 to 12.28] — Odds for travel in the prior 3 months as a risk factor for Heavy drinking (>14 and >21 drinks/week for women and men respectively) in the past 30 days
Statistical Analysis 7: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 3.63, 95% CI 2-sided [2.02 to 6.50] — Adjusted odds for travel in the prior 3 months as a risk factor for Drank until blacked out in the past 30 days
Statistical Analysis 8: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p = 0.04, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.33 to 0.93] — Adjusted odds for travel in the prior 3 months as a risk factor for Injected daily, past 30 days
Statistical Analysis 9: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence intervals for travel as a risk factor for each behavior; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.37 to 3.40] — Adjusted odds for travel in the prior 3 months as a risk factor for Median number of injected partners >= 5 in the past 30 days
Statistical Analysis 10: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence interval for travel in the prior 3 months as a risk factor for having Lent a needle/syringe in the past 30 days; Test type: Superiority or Other; p = 0.19, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.81 to 1.97] — Adjusted odds for travel in prior 3 months as a risk factor for having Lent a needle/syringe in the past 30 days
Statistical Analysis 11: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds ratio with 95 % confidence interval for travel in prior 3 months as a risk factor for having injected with someone else's used needle/syringe in the past 30 days; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.01 to 2.55] — Adjusted odds for travel in prior 3 months as a risk factor for having Injected with someone else's used needle/syringe in the past 30 days
Statistical Analysis 12: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence interval for travel in the prior 3 months as a risk factor for having Pooled money to buy drugs in the past 30 days; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 3.07, 95% CI 2-sided [1.79 to 5.27] — Adjusted odds for travel in prior 3 months as a risk factor for having Pooled money to buy drugs in the past 30 days
Statistical Analysis 13: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds ratios with 95% confidence interval for travel in prior 3 months as risk factor for risk behaviors; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.34 to 3.32] — Adjusted odds for travel in prior 3 months as a risk factor for having Shared cooker/spook to prepare drugs in the past 30 days
Statistical Analysis 14: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95 % confidence interval for travel as a risk factor for risk behaviors; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.19 to 2.95] — Adjusted odds for travel in prior 3 months as a risk factor for having used Backloaded Syringe in the past 30 days
Statistical Analysis 15: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds with 95% confidence interval for travel in prior 3 months as a risk factor for risk behavior in past 30 days; Test type: Superiority or Other; p = 0.13, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.83 to 2.10] — Adjusted odds for travel in prior 3 months as a risk factor for having done Someone's "rinse" in the past 30 days
Statistical Analysis 16: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds ratios and 95% confidence intervals for travel in prior 3 months as a risk factor for risk behaviors in past 30 days; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.40 to 3.49] — Adjusted odds for travel in prior 3 months as a risk factor for Median number of sexual partners >=2 in the past 30 days
Statistical Analysis 17: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds and 95% confidence interval for travel in prior 3 months as a risk factor for risk behaviors in past 30 days; Test type: Superiority or Other; p = 0.86, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.45 to 1.85] — Adjusted odds for travel in prior 3 months as a risk factor for having Traded sex for money or drugs in the past 30 days
Statistical Analysis 18: Comparison: Traveled in the Prior 3 Months vs Did Not Travel in the Prior 3 Months; Adjusted odds and 95% confidence interval for travel in prior 3 months as a risk factor for engaging in risk behavior during the past 30 days; Test type: Superiority or Other; p = 0.73, Regression, Logistic; Odds ratios adjusted for age, race, sex, years injecting; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.59 to 2.02] — Adjusted odds for travel in prior 3 months as a risk factor for condom use >90% (if sexually active)

4. Secondary Outcome: HIV Vaccine Trial Willingness
Description: We assessed knowledge about vaccine trials and willingness to participate in preventive HIV vaccine trials by asking the question: "How willing would you be to join a study of a vaccine to prevent HIV infection, if the study were to start tomorrow?". Willingness was measured on a 4-point response scale, ranging from 1 (Definitely not willing) to 4 (Definitely willing).
Time Frame: Baseline
Population: Per the Participant Flow, 409 participants in the cross-sectional study had complete and valid baseline data
Measure: Number; unit: Participants
Groups:
- Cross-sectional Study Participants: Participants enrolled in the pre-randomization cross-sectional screening study completed a 60-minute survey, received client-centered risk reduction counseling, and underwent phlebotomy for viral testing. Participants were invited to return one week later for viral testing results, counseling, referrals, and subsequent enrollment in the vaccine adherence cohort study, if eligible.
Arm/Group | Cross-sectional Study Participants
Number analyzed (Participants) | 409
Participants
  1=Definitely not willing | 24
  2=Probably not willing | 68
  3=Probably willing | 170
  4=Definitely willing | 147

5. Secondary Outcome: HIV Vaccine Trial Knowledge
Description: Participants were asked if they agreed or disagreed with or were unsure of each of eight statements about HIV vaccine trial concepts from the HIV Network for Prevention Trials (HIVNET).
  1. Preventive HIV vaccine studies enroll people who are HIV-positive and HIV-negative.
  2. Some participants in HIV vaccine studies will get a real vaccine, and some will get a placebo (an inactive substance).
  3. Only vaccines known to be at least 50% effective at preventing HIV are tested in HIV vaccine studies.
  4. Once a large scale HIV vaccine study begins, we can be sure the vaccine is completely safe.
  5. Participants are told whether they got the HIV vaccine or the placebo at the end of HIV vaccine studies.
  6. HIV vaccines will never affect a person's HIV test results.
  7. An HIV vaccine can infect a person with HIV disease.
  8. People in vaccine studies know whether or not they got the placebo because only the vaccines cause side effects.
Time Frame: Baseline
Population: Per the Participant Flow, 409 participants in the cross-sectional study had complete and valid baseline data
Measure: Number; unit: Participants
Groups:
- Screening Study Participants: Participants enrolled in the pre-randomization cross-sectional screening study completed a 60-minute survey, received client-centered risk reduction counseling, and underwent phlebotomy for viral testing. Participants were invited to return one week later for viral testing results, counseling, referrals, and subsequent enrollment in the vaccine adherence cohort study, if eligible.
Arm/Group | Screening Study Participants
Number analyzed (Participants) | 409
Participants
  5-8 Correct answers | 94
  0-4 Correct answers | 315

ADVERSE EVENTS:
Time Frame: 12 months
Description: Participants were observed for 10-15 minutes following each vaccination and instructed to contact the clinic if any adverse event was experienced.
Arm/Group | AIC Only | AIC + Outreach | SEP Only | SEP + Outreach
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/43 | 0/36 | 0/41
Other Adverse Events (participants affected / at risk) | 0/47 | 0/43 | 0/36 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No